CLINICAL TRIAL: NCT05848258
Title: An Adaptive Phase 2a/2b, Randomized, Double-Blind, Placebo-Controlled Study of LY3871801 in Adult Participants With Moderately-to-Severely Active Rheumatoid Arthritis
Brief Title: An Adaptive Phase 2a/2b Study of LY3871801 in Adult Participants With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18516; J3P-MC-FTAF (Other: Eli Lilly and Company); 2022-502994-40-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3871801 Phase 2a (Experimental): Participants will receive LY3871801 administered orally.
  Interventions: Drug: LY3871801
- Placebo Phase 2a (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo
- LY3871801 Dose 1 Phase 2b (Experimental): Participants will receive LY3871801 administered orally.
  Interventions: Drug: LY3871801
- LY3871801 Dose 2 Phase 2b (Experimental): Participants will receive LY3871801 administered orally.
  Interventions: Drug: LY3871801
- LY3871801 Dose 3 Phase 2b (Experimental): Participants will receive LY3871801 administered orally.
  Interventions: Drug: LY3871801
- Placebo Phase 2b (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3871801 — Administered orally
  Arms: LY3871801 Dose 1 Phase 2b; LY3871801 Dose 2 Phase 2b; LY3871801 Dose 3 Phase 2b; LY3871801 Phase 2a
Drug: Placebo — Administered orally
  Arms: Placebo Phase 2a; Placebo Phase 2b

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of LY3871801 in adult participants with active moderately-to-severe rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset RA for at least 3 months prior to screening as defined by the 2010 ACR/European League Against Rheumatism (EULAR) classification criteria.
* Have moderately-to-severely active RA at screening and baseline, defined by the presence of

  * ≥6 swollen joints based on 66 joint count, and
  * ≥6 tender joints based on 68 joint count.
* Have had a history of failure (an inadequate response, intolerance, or loss of response) to at least 1 conventional synthetic disease modifying anti rheumatic drug (csDMARD) and either 1 biologic (bDMARD), or targeted synthetic (tsDMARD) treatment.

Exclusion Criteria:

* Have Class IV RA according to ACR revised criteria
* Have presence of 1 or more significant concurrent medical conditions per investigator judgment, including but not limited to

  * poorly controlled diabetes or hypertension
  * chronic kidney disease stage IIIa or IIIb, IV, or V
  * symptomatic heart failure according to New York Heart Association class II, III, or IV
  * myocardial infarction,unstable angina pectoris, stroke, or transient ischemic attack within the past 12 months before randomization
  * severe chronic pulmonary disease, for example, requiring oxygen therapy
  * major chronic inflammatory disease or connective tissue disease other than RA, including but not limited to

    * systemic lupus erythematosus
    * psoriatic arthritis
    * axial spondyloarthritis,including ankylosing spondylitis and non-radiographic axial spondyloarthritis
    * reactive arthritis
    * gout
    * scleroderma
    * polymyositis
    * dermatomyositis
    * active fibromyalgia, or
    * multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Phase 2a: Change from Baseline in Disease Activity Score - high-sensitivity C-reactive protein (DAS28-hsCRP) | Baseline, Week 12
Phase 2b: Percentage of Participants Achieving American College of Rheumatology (ACR)50 | Baseline to Week 12

SECONDARY OUTCOMES:
Phase 2a: Percentage of Participants Achieving ACR20/50/70 | Baseline to Week 12
Phase 2b: Change from Baseline in DAS28-hsCRP | Baseline, Week 12
Phase 2b: Percentage of Participants Achieving ACR20/70 | Week 12
Change from Baseline in Simplified Disease Activity Index (SDAI) | Baseline, Week 12
Change from Baseline in Clinical Disease Activity Index (CDAI) | Baseline, Week 12
Change from Baseline in ACR Core Set Values 68 Tender Joint Counts | Baseline, Week 12
Change from Baseline in ACR Core Set Values 66 Swollen Joint Counts | Baseline, Week 12
Change from Baseline in ACR Core Set Values Physician's Global Assessment of Disease Activity (PhGADA) Visual Analog Scale (VAS) | Baseline, Week 12
Change from Baseline in ACR Core Set Values Patient's Global Assessment of Disease Activity (PaGADA) VAS | Baseline, Week 12
Change from Baseline for Participant's Assessment of Arthritis Pain (VAS) | Baseline, Week 12
Change from Baseline for Participant's Assessment of Physical Function Using Health Assessment Questionnaire-Disability Index (HAQ-DI) | Baseline, Week 12
Change from Baseline the Duration and Severity of Morning Joint Stiffness | Baseline, Week 12
Change from Baseline for Short Form-36 (SF-36) Physical Component Summary Score | Baseline, Week 12
Change from Baseline for SF-36 Mental Component Summary Score | Baseline, Week 12
Pharmacokinetics (PK) Trough Plasma Concentrations of LY3871801 | Baseline through Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (57):
- United States (12):
  - Newport Huntington Medical Group, Huntington Beach, California
  - Integrity Clinical Research, Doral, Florida
  - Advanced Clinical Research of Orlando - Ocoee, Ocoee, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Conquest Research, Winter Park, Florida
  - Willow Rheumatology and Wellness PLLC, Willowbrook, Illinois
  - Accurate Clinical Research, Inc, Lake Charles, Louisiana
  - Joseph S. and Diane H. Steinberg Ambulatory Care Center, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Accellacare - Salisbury, Salisbury, North Carolina
  - Accurate Clinical Research, Inc, Houston, Texas
  - Overlake Arthritis and Osteoporosis Center, Bellevue, Washington
- Argentina (5):
  - CIPREC, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - CENUDIAB, Buenos Aires
  - Medicina Reumatológica, San Fernando
  - Instituto de Alta Complejidad San Isidro, San Isidro
- Medical Plus, Uherské Hradiště, Czechia
- France (7):
  - CHD Vendee, La Roche-sur-Yon
  - CHU Montpellier Lapeyronie Hospital, Montpellier
  - CHU de Nice, Nice
  - Centre Hospitalier Regional D'Orleans, Orléans
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Centre Hospitalier Universitaire de Reims - l'Hôpital Maison Blanche, Reims
  - CHU Strasbourg-Hautepierre, Strasbourg
- Germany (2):
  - Universitaetsklinikum Koeln, Cologne
  - HRF II - Hamburger Rheuma Forschungszentrum II MVZ für Rheumatologie und Autoimmunmedizin Hamburg GmbH / -T, Hamburg
- Hungary (8):
  - Revita Clinic, Budapest
  - Clinexpert Kft., Budapest
  - Óbudai Egészségügyi Centrum, Budapest
  - CRU Hungary Kft., Encs
  - Vásárhelyi Sárkányfű KFT, Hódmezővásárhely
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - Regia Med Kft, Székesfehérvár
  - Vital Medical Center, Veszprém
- India (7):
  - Avron Hospitals, Ahmedabad
  - Sushruta Multispeciality Hospital & Research Centre, Hubli
  - Government Medical College And Hospital - Nagpur, Nagpur
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - Grant Medical Foundation - Ruby Hall Clinic, Pune
  - Medipoint Hospitals Pvt. Ltd., Pune
  - All India Institute of Medical Sciences, Raipur
- Mexico (9):
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
  - Hospital Aranda de La Parra, León
  - Biológicos Especializados, Mexico City
  - Kohler and Milstein Research S.A. de C.V., Mérida
  - Medical Care and Research SA de CV, Mérida
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - Cicmex Centro de Investigación Clínica de México, Morelia
  - Centro de Atención e Investigación Cardiovascular del Potosí, San Luis Potosí City
  - CIMAB SA de CV, Torreón
- Poland (4):
  - Nova Reuma Domyslawska i Rusilowicz Spolka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok
  - Nzoz Bif-Med, Bytom
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
- United Kingdom (2):
  - Hull Royal Infirmary, Hull
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: An Adaptive Phase 2a/2b Study of LY3871801 in Adult Participants With Rheumatoid Arthritis — https://trials.lilly.com/en-US/trial/401857